CLINICAL TRIAL: NCT04184843
Title: Development and Evaluation of iWalk: A Guide to Facilitate Evidence-informed Assessment of Walking After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Dalhousie University (Other); University Health Network, Toronto (Other); Nova Scotia Health Authority (Other); McMaster University (Other); CorHealth Ontario (Other); Drexel University (Other); Sunnybrook Health Sciences Centre (Other); Sinai Health System (Other); Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Dr. Nancy Salbach, Associate Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KAL322155
Record Dates: First submitted 2019-11-08; First posted 2019-12-04 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iWalk Toolkit (Experimental): Intervention period: 5 months
  Intervention:
  1. A toolkit consisting of 3 components: an educational guide, a smartphone app, and an educational video.
  2. Access to a clinical expert by email or phone
  Interventions: Other: iWalk Toolkit

INTERVENTIONS:
Other: iWalk Toolkit — Intervention period: 5 months
  Intervention:
  1. A toolkit consisting of 3 components: an educational guide, a smartphone app, and an educational video.
  2. Access to a clinical expert by email or phone

SUMMARY:
Stroke remains a major health concern and the second highest cause of disability worldwide. After experiencing a stroke, many people lose the ability to walk independently. As a result, people with stroke require intensive rehabilitation services, spend the majority of their time in physical therapy on retraining walking, and cite recovery of walking as a primary rehabilitation goal. Assessment of walking using reliable and valid tools is a recommended practice in stroke rehabilitation guidelines in Canada, the United States, Australia, and The Netherlands. The 10-metre walk test (10mWT) and the 6-minute walk test (6MWT) are highly recommended in guidelines and by professional organizations for the clinical evaluation of walking across the care continuum. For the 10mWT, the time to traverse the middle 10 metres of a 14-metre walkway at a comfortable pace is used to compute comfortable walking speed. For the 6MWT, the maximum distance achieved walking back and forth along a 30-metre walkway in six minutes is documented.

To facilitate physical therapists' (PTs') use of an evidence-informed approach to administering these walking tests post-stroke in an acute care, inpatient rehabilitation, or outpatient rehabilitation setting, the iWalk Toolkit, a theory-based toolkit, was developed. This Toolkit consists of an educational guide, a smartphone app, and an educational video.

In this mixed methods study, PTs across multiple sites were evaluated before and after a 5-month intervention involving the implementation of the iWalk Toolkit. Objectives of this study were: (1) to determine the nature and extent to which PTs across the care continuum uptake/use information in a theory-based toolkit designed to guide use of the 10-metre and 6-minute walk tests post-stroke for initial assessment, goal setting, education, treatment selection and monitoring change; and (2) to describe PTs' perceptions of the features of the guide, the provider and the setting that facilitated or prevented walk test administration and use of test scores for initial assessment, prognosis, goal setting, treatment selection and monitoring change.

ELIGIBILITY:
Inclusion Criteria:

* Physical therapists working in hospitals providing acute care, in-patient rehabilitation, or outpatient rehabilitation services for people with stroke
* Physical therapists registered with the provincial regulatory body
* Physical therapists who provided walking rehabilitation to 10 or more patients with stroke per year
* Individuals in a professional leader (PL) or professional practice leader (PPL) role defined as an individual who was responsible for facilitating and advancing evidence-based physical therapy practice and ensuring that professional practice standards were met.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change in the percentage of ambulatory patients post-stroke for which physical therapists have documented administration of walk tests in the health record at least once during the patient's hospital stay or physical therapy treatment | Change from baseline to 5 months
  Data collected from patient health records pre- and post-intervention

SECONDARY OUTCOMES:
Change in the percentage of physical therapists in the action or maintenance stage determined using the 26-item self-report Clinician Readiness for Measuring Outcomes Scale. | Change from baseline to 5 months
  Data collected from pre- and post-intervention online questionnaire.
Change in the mean self-efficacy rating on an 11-point ordinal scale ranging from 0% (no confidence) to 100% (completely confident) for physical therapists performing 12 unique walk test practices. | Change from baseline to 5 months
  Data collected from pre- and post-intervention online questionnaire.
Median score from 1 (inadequate) to 5 (excellent) for each domain (engagement, functionality, aesthetics, and information quality) on the Mobile App Rating Scale (MARS). | At 5 months
  Data collected from post-intervention online questionnaire.
Percentage of therapists who attended each learning session, reviewed each iWalk guide module and the video, practiced each walk test with colleagues, completed learning activities outlined in the guide, and used the app in clinical or various practices. | At 5 months
  Participants indicated extent to which app was used in clinical practice (1, 2, 3, 4, or 5 months), and for various practices (none/little of the time, some of the time, or most/all of the time).
  Data collected from post-intervention online questionnaire.
Physical therapists' perceptions of the features of the guide, the provider and the setting that facilitated or prevented walk test administration and use of test scores | Up to 8 months
  Data collected from face-to-face or telephone interviews and focus groups held with participants post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Salbach, PhD, Principal Investigator — University of Toronto

REFERENCES:
- [Derived] Salbach NM, MacKay-Lyons M, Howe JA, McDonald A, Solomon P, Bayley MT, McEwen S, Nelson M, Bulmer B, Lovasi GS. Assessment of Walking Speed and Distance Post-Stroke Increases After Providing a Theory-Based Toolkit. J Neurol Phys Ther. 2022 Oct 1;46(4):251-259. doi: 10.1097/NPT.0000000000000406. Epub 2022 Jun 7. PMID 35671402